CLINICAL TRIAL: NCT03681613
Title: Randomized Controlled Trial of Exercise Therapy in Combination With Central Nervous System-targeted Treatment Compared With Exercise Therapy Alone for Treatment of People With Knee Osteoarthritis
Brief Title: Exercise Therapy in Combination With Central Nervous System-targeted Treatment for Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Enrique Lluch Girbés, PhD Professor, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H1526892955402
Record Dates: First submitted 2018-09-18; First posted 2018-09-24 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2023-06

CONDITIONS: Osteoarthritis; Osteo Arthritis Knee
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Therapy With CNS Treatment (Experimental): NEMEX program combined with a CNS-focused protocol
  Interventions: Other: NEMEX program combined with a CNS-focused protocol
- Exercise Therapy alone (Experimental): NEMEX program alone
  Interventions: Other: NEMEX program

INTERVENTIONS:
Other: NEMEX program combined with a CNS-focused protocol — The NEMEX program will consist of 12-weeks of individualized and supervised exercise sessions applied twice weekly (n=24 sessions). Each exercise session will last approximately 60minutes and include three parts: warming up, a circuit program and cooling down.
  The CNS-targeted treatment will consist of 12-week individualized and supervised sessions applied once weekly. Each training session will last approximately 30 minutes and include three parts, which are further explained below: 1) discussion of the participant's knee pain experience from a pain neuroscience perspective, 2) graded SDT and 3) GMI training.
  Other Names: Graded Motor Imagery; Sensory Discrimination Training; NEMEX program
  Arms: Exercise Therapy With CNS Treatment
Other: NEMEX program — The NEMEX program will consist of 12-weeks of individualized and supervised exercise sessions applied twice weekly (n=24 sessions). Each exercise session will last approximately 60minutes and include three parts: warming up, a circuit program and cooling down.
  Arms: Exercise Therapy alone

SUMMARY:
The aim of this study is to investigate if exercise therapy comprising the NEMEX program in combination with a CNS-targeted treatment using GMI and SDT is superior to exercise therapy alone in improving self-reported pain, function, quality of life and objective measures related to hyperexcitability of the CNS (e.g. central sensitization) in people with KOA.

DETAILED DESCRIPTION:
Participants will be randomized to one of two treatments initiated after randomization: the NEMEX program combined with a CNS-focused protocol or the NEMEX program alone.

The NEMEX program will consist of 12-weeks of individualized and supervised exercise sessions applied twice weekly (n=24 sessions). Each exercise session will last approximately 60minutes and include three parts: warming up, a circuit program and cooling down.

The CNS-targeted treatment will consist of 12-week individualized and supervised sessions applied twice weekly. Each training session will last approximately 30 minutes and include three parts, which are further explained below: 1) discussion of the participant's knee pain experience from a pain neuroscience perspective, 2) graded SDT and 3) GMI training.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic and radiographically-confirmed tibiofemoral KOA (e.g. Kellgren-Lawrence ≥2, scored by an orthopaedic surgeon, not scheduled for total knee replacement [decision among other factors based on pain, function and radiographic severity.
* Diagnosis of KOA according to the EULAR classification criteria: adults aged >40 years with usage-related knee pain, only short-lived (<30min) morning stiffness, functional limitation (based on yes/no to the following question: Is your functional level reduced as compared to before your knee symptoms first started?) and one or more typical examination findings (crepitus, restricted movement, bony enlargement). The presence of this cluster correctly diagnosed 99% of cases with KOA.

Exclusion Criteria:

* Less than mild functional limitations (a score above 75 on a 0-100 worst to best scale in the Spanish version of the self-report questionnaire Knee injury and Osteoarthritis Outcome Score (KOOS)4 defined as the average score for the subscale scores for pain, symptoms, activities of daily living (ADL) and quality of life (QOL).
* Previous knee replacement or any other lower limb surgery in the affected knee within the previous 3 months.
* Fracture of the affected extremity within the previous 6 months.
* Initiation of opioid analgesia or any form of injection (i.e. corticosteroid, hyaluronic acid, platelet-rich plasma) for knee pain within the previous 30 days.
* Physical impairments unrelated to the knee that would prevent safe participation in exercise.
* Any comorbidity that prevents from participating in the interventions (e.g.uncontrolled hypertension, moderate to high risk for cardiac complications)
* Any skin or medical condition preventing tactile stimulation on the knee.
* Inability to comprehend and complete study assessments or comply with study instructions (e.g. illiteracy, cognitive or visual impairments).
* Inability to a priori attend or complete the proposed course of intervention and follow-up schedule.

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2019-01-07 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
The Knee injury and Osteoarthritis Outcome Score subscales (KOOS4) | baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  The primary outcome is the between-group difference in change in the mean score on four Knee Injury and Osteoarthritis Outcome Score (KOOS) subscales, covering pain, symptoms, activities of daily living, and quality of life (KOOS4).
  The four patient-relevant subscales of KOOS are scored separately: Pain (9 items); Symptoms (7 items); ADL Function (17 items); Quality of Life (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the four scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.

SECONDARY OUTCOMES:
The Knee injury and Osteoarthritis Outcome Score (KOOS) | baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  The KOOS is a knee-specific instrument, developed to assess the patients' opinion about their knee and associated problems. It holds 42 items in 5 separately scored subscales; Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL).
  The scores on all five patient-relevant subscales of KOOS are scored separately: Pain (9 items); Symptoms (7 items); ADL Function (17 items); Sport and Recreation Function (5 items); Quality of Life (4 items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Pain intensity: NRS | baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  Participants will be presented with four numerical rating scales anchored with 0 ("no pain") and 10 ("pain as bad as you can imagine"): 1) rating the most intense pain over the last week, 2) rating the least intense pain over the last week, 3) rating the average pain intensity over the last week, and 4) rating the pain right now. The scores will be averaged to calculate a final pain intensity score out of 10
Sensitivity to physical activity | baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  Participants will be asked to rate their level of knee discomfort before, during, and after the 30-s chair-stand test in accordance with previous studies (Wideman et al., 2014). Knee discomfort will be ranked three times on a verbal rating scale that ranged from 0 (no discomfort) to 100 (extreme discomfort), once immediately before the task, once during the middle and once at the end of the task. An index of sensitivity to physical activity (SPA) will be calculated by subtracting participants' first rating from their last rating.
General health | baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  General health will be assessed using the Spanish version of the EuroQol Group 5-Dimension (EQ-5D-5L) self-reported questionnaire. EQ-5D-5L is a questionnaire with 5 dimensions (mobility, self-care, usual activities, pain/ discomfort, and anxiety/depression) and 5 levels in each dimension (no problems, slight, moderate, severe, and un- able or extreme). Each health state is usually represented using a 5-digit number (profile) where 11111 indicates perfect health and 55555 the worst health state or pits state.
Cortical representation | baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  The two-point discrimination (TPD) threshold is considered a clinical signature of cortical representation primary somatosensory representation. The TPD threshold will be measured using a mechanical sliding calliper (Duratech TA-2081, precision = 1 mm) in the vertical direction on the affected knee using suprathreshold (but non-noxious stimuli) and following an established protocol.
Pressure pain thresholds | baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  A standardized protocol for evaluating PPTs will be used. Two test sites in the peripatellar region (3 cm medial and lateral to the midpoint of the medial and lateral edge of patella, respectively) and one distant site on the ipsilateral trapezius muscle (midpoint between spinous process of C7 and lateral border of acromion) will be selected for measurement. The PPT will be measured using an analogue Fisher algometer (Force Dial model FDK 40) with a surface area of 1cm2. The algometer probe tip was applied perpendicular to the skin at a rate of 1kg/cm2/s until the first onset of pain. Three measures were performed on each site with a 30 s interstimulus interval between each measurement and the mean was taken for analysis.
Central Sensitization Inventory | baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  To identify key symptoms associated with augmented central pain processing mechanisms (e.g.central sensitization), the Spanish version of the Central Sensitization Inventory will be used (Cuesta-Vargas et al., 2016). The CSI provides reliable and valid data that quantify the severity of several symptoms of CS (Scerbo et al., 2017).
Conditioned Pain Modulation | baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  Conditioned pain modulation (CPM) was tested using the upper extremity submaximal effort tourniquet test. Three trials of PPT measures at the two sites in the peripatellar region (medial and lateral to the midpoint of the medial and lateral edge of patella) were taken immediately following deflation.
Number of participants with adverse events and number of adverse events | During follow-up
  Adverse events (AE) and serious adverse events (SAEs) will be recorded at all follow-ups by asking patients about potential AEs using open-probe questioning to ensure that all AEs are recorded. In addition, the physiotherapist will record any adverse events that the patient experiences or talks about during treatment.
Global perceived effect, patient acceptable symptom state and treatment failure | 12 months after initiating the treatment
  Global perceived effect will be assessed with the question: "How are your knee problems now compared with before you entered this study?" This question will be answered on a Likert scale ranging from 1 ("very much improved") to 7 ("very much worse").
  Satisfaction with current knee function will be evaluated by the following question: "When you think of your knee function, will you consider your current condition as satisfying?"
Compliance, exercise level/intensity and other treatments received during the study | Up to 12 weeks
  Compliance with treatment sessions will be monitored by the supervising physiotherapists using an individual treatment diary where the number of sessions, progression of the exercises (e.g. level of difficulty at which all specific exercises are performed each session), time of day and duration of each clinic session will be recorded.
Knee flexor and extensor strength | Baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  Isometric knee flexor and extensor strength testing with modified hand-held dynamometry will be performed.
Number of chair stands in 30 seconds | Baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  As performance-based tests of physical function, the number of chair stands will be assessed. These tests have been recommended as performance-based tests of physical function representing typical activities relevant to individuals diagnosed with KOA.
40 m fast-paced walk test | Baseline, post-intervention (after 12 weeks) and 6 and 12 months after initiating the treatment
  As performance-based tests of physical function, the 40 m fast-paced walk test will be assessed in seconds. These tests have been recommended as performance-based tests of physical function representing typical activities relevant to individuals diagnosed with KOA.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Lluch Girbés, PhD, Study Director — University of Valencia; Søren Thorgaard Skou, PhD, Study Chair — University of Southern Denmark; Javier Peral Pérez, PhD student, Principal Investigator — University of Alcalá
Locations (1):
- University of Valencia, Valencia, Spain

REFERENCES:
- [Background] Abaei M, Sagar DR, Stockley EG, Spicer CH, Prior M, Chapman V, Auer DP. Neural correlates of hyperalgesia in the monosodium iodoacetate model of osteoarthritis pain. Mol Pain. 2016 Apr 11;12:1744806916642445. doi: 10.1177/1744806916642445. Print 2016. PMID 27068285
- [Background] Ageberg E, Link A, Roos EM. Feasibility of neuromuscular training in patients with severe hip or knee OA: the individualized goal-based NEMEX-TJR training program. BMC Musculoskelet Disord. 2010 Jun 17;11:126. doi: 10.1186/1471-2474-11-126. PMID 20565735
- [Background] Ageberg E, Nilsdotter A, Kosek E, Roos EM. Effects of neuromuscular training (NEMEX-TJR) on patient-reported outcomes and physical function in severe primary hip or knee osteoarthritis: a controlled before-and-after study. BMC Musculoskelet Disord. 2013 Aug 8;14:232. doi: 10.1186/1471-2474-14-232. PMID 23924144
- [Background] Ageberg E, Roos EM. Neuromuscular exercise as treatment of degenerative knee disease. Exerc Sport Sci Rev. 2015 Jan;43(1):14-22. doi: 10.1249/JES.0000000000000030. PMID 25390299
- [Background] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Background] Arendt-Nielsen L, Skou ST, Nielsen TA, Petersen KK. Altered Central Sensitization and Pain Modulation in the CNS in Chronic Joint Pain. Curr Osteoporos Rep. 2015 Aug;13(4):225-34. doi: 10.1007/s11914-015-0276-x. PMID 26026770
- [Background] Arendt-Nielsen L. Joint pain: more to it than just structural damage? Pain. 2017 Apr;158 Suppl 1:S66-S73. doi: 10.1097/j.pain.0000000000000812. No abstract available. PMID 28151834
- [Background] Arendt-Nielsen L, Morlion B, Perrot S, Dahan A, Dickenson A, Kress HG, Wells C, Bouhassira D, Drewes AM. Assessment and manifestation of central sensitisation across different chronic pain conditions. Eur J Pain. 2018 Feb;22(2):216-241. doi: 10.1002/ejp.1140. Epub 2017 Nov 5. PMID 29105941
- [Background] Baliki MN, Schnitzer TJ, Bauer WR, Apkarian AV. Brain morphological signatures for chronic pain. PLoS One. 2011;6(10):e26010. doi: 10.1371/journal.pone.0026010. Epub 2011 Oct 13. PMID 22022493
- [Background] Bartholdy C, Juhl C, Christensen R, Lund H, Zhang W, Henriksen M. The role of muscle strengthening in exercise therapy for knee osteoarthritis: A systematic review and meta-regression analysis of randomized trials. Semin Arthritis Rheum. 2017 Aug;47(1):9-21. doi: 10.1016/j.semarthrit.2017.03.007. Epub 2017 Mar 18. PMID 28438380
- [Background] Bennell KL, Hunt MA, Wrigley TV, Lim BW, Hinman RS. Role of muscle in the genesis and management of knee osteoarthritis. Rheum Dis Clin North Am. 2008 Aug;34(3):731-54. doi: 10.1016/j.rdc.2008.05.005. PMID 18687280
- [Background] Bowering KJ, O'Connell NE, Tabor A, Catley MJ, Leake HB, Moseley GL, Stanton TR. The effects of graded motor imagery and its components on chronic pain: a systematic review and meta-analysis. J Pain. 2013 Jan;14(1):3-13. doi: 10.1016/j.jpain.2012.09.007. Epub 2012 Nov 15. PMID 23158879
- [Background] Carr AJ, Robertsson O, Graves S, Price AJ, Arden NK, Judge A, Beard DJ. Knee replacement. Lancet. 2012 Apr 7;379(9823):1331-40. doi: 10.1016/S0140-6736(11)60752-6. Epub 2012 Mar 6. PMID 22398175
- [Background] Catley MJ, Tabor A, Wand BM, Moseley GL. Assessing tactile acuity in rheumatology and musculoskeletal medicine--how reliable are two-point discrimination tests at the neck, hand, back and foot? Rheumatology (Oxford). 2013 Aug;52(8):1454-61. doi: 10.1093/rheumatology/ket140. Epub 2013 Apr 22. PMID 23611918
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Chang AH, Lee SJ, Zhao H, Ren Y, Zhang LQ. Impaired varus-valgus proprioception and neuromuscular stabilization in medial knee osteoarthritis. J Biomech. 2014 Jan 22;47(2):360-6. doi: 10.1016/j.jbiomech.2013.11.024. Epub 2013 Nov 25. PMID 24321442
- [Background] Chang WJ, Bennell KL, Hodges PW, Hinman RS, Young CL, Buscemi V, Liston MB, Schabrun SM. Addition of transcranial direct current stimulation to quadriceps strengthening exercise in knee osteoarthritis: A pilot randomised controlled trial. PLoS One. 2017 Jun 30;12(6):e0180328. doi: 10.1371/journal.pone.0180328. eCollection 2017. PMID 28665989
- [Background] Clausen B, Holsgaard-Larsen A, Roos EM. An 8-Week Neuromuscular Exercise Program for Patients With Mild to Moderate Knee Osteoarthritis: A Case Series Drawn From a Registered Clinical Trial. J Athl Train. 2017 Jun 2;52(6):592-605. doi: 10.4085/1062-6050-52.5.06. PMID 28653869
- [Background] Courtney CA, Steffen AD, Fernandez-de-Las-Penas C, Kim J, Chmell SJ. Joint Mobilization Enhances Mechanisms of Conditioned Pain Modulation in Individuals With Osteoarthritis of the Knee. J Orthop Sports Phys Ther. 2016 Mar;46(3):168-76. doi: 10.2519/jospt.2016.6259. Epub 2016 Jan 1. PMID 26721229
- [Background] Cuesta-Vargas AI, Roldan-Jimenez C, Neblett R, Gatchel RJ. Cross-cultural adaptation and validity of the Spanish central sensitization inventory. Springerplus. 2016 Oct 21;5(1):1837. doi: 10.1186/s40064-016-3515-4. eCollection 2016. PMID 27818875
- [Background] Daffada PJ, Walsh N, McCabe CS, Palmer S. The impact of cortical remapping interventions on pain and disability in chronic low back pain: a systematic review. Physiotherapy. 2015 Mar;101(1):25-33. doi: 10.1016/j.physio.2014.07.002. Epub 2014 Aug 1. PMID 25442672
- [Background] Dobson F, Hinman RS, Roos EM, Abbott JH, Stratford P, Davis AM, Buchbinder R, Snyder-Mackler L, Henrotin Y, Thumboo J, Hansen P, Bennell KL. OARSI recommended performance-based tests to assess physical function in people diagnosed with hip or knee osteoarthritis. Osteoarthritis Cartilage. 2013 Aug;21(8):1042-52. doi: 10.1016/j.joca.2013.05.002. Epub 2013 May 13. PMID 23680877
- [Background] Escobar A, Quintana JM, Bilbao A, Azkarate J, Guenaga JI. Validation of the Spanish version of the WOMAC questionnaire for patients with hip or knee osteoarthritis. Western Ontario and McMaster Universities Osteoarthritis Index. Clin Rheumatol. 2002 Nov;21(6):466-71. doi: 10.1007/s100670200117. PMID 12447629
- [Background] Fernandes L, Hagen KB, Bijlsma JW, Andreassen O, Christensen P, Conaghan PG, Doherty M, Geenen R, Hammond A, Kjeken I, Lohmander LS, Lund H, Mallen CD, Nava T, Oliver S, Pavelka K, Pitsillidou I, da Silva JA, de la Torre J, Zanoli G, Vliet Vlieland TP; European League Against Rheumatism (EULAR). EULAR recommendations for the non-pharmacological core management of hip and knee osteoarthritis. Ann Rheum Dis. 2013 Jul;72(7):1125-35. doi: 10.1136/annrheumdis-2012-202745. Epub 2013 Apr 17. PMID 23595142
- [Background] Fingleton C, Smart K, Moloney N, Fullen BM, Doody C. Pain sensitization in people with knee osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Jul;23(7):1043-56. doi: 10.1016/j.joca.2015.02.163. Epub 2015 Mar 5. PMID 25749012
- [Background] Fitzgerald GK, Piva SR, Irrgang JJ. Reports of joint instability in knee osteoarthritis: its prevalence and relationship to physical function. Arthritis Rheum. 2004 Dec 15;51(6):941-6. doi: 10.1002/art.20825. PMID 15593258
- [Background] Flor H. Cortical reorganisation and chronic pain: implications for rehabilitation. J Rehabil Med. 2003 May;(41 Suppl):66-72. doi: 10.1080/16501960310010179. PMID 12817660
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Harvey AK, Taylor AM, Wise RG. Imaging pain in arthritis: advances in structural and functional neuroimaging. Curr Pain Headache Rep. 2012 Dec;16(6):492-501. doi: 10.1007/s11916-012-0297-4. PMID 23011761
- [Background] Hochberg MC, Altman RD, April KT, Benkhalti M, Guyatt G, McGowan J, Towheed T, Welch V, Wells G, Tugwell P; American College of Rheumatology. American College of Rheumatology 2012 recommendations for the use of nonpharmacologic and pharmacologic therapies in osteoarthritis of the hand, hip, and knee. Arthritis Care Res (Hoboken). 2012 Apr;64(4):465-74. doi: 10.1002/acr.21596. PMID 22563589
- [Background] Huber EO, Roos EM, Meichtry A, de Bie RA, Bischoff-Ferrari HA. Effect of preoperative neuromuscular training (NEMEX-TJR) on functional outcome after total knee replacement: an assessor-blinded randomized controlled trial. BMC Musculoskelet Disord. 2015 Apr 25;16:101. doi: 10.1186/s12891-015-0556-8. PMID 25925404
- [Background] Ingelsrud LH, Granan LP, Terwee CB, Engebretsen L, Roos EM. Proportion of Patients Reporting Acceptable Symptoms or Treatment Failure and Their Associated KOOS Values at 6 to 24 Months After Anterior Cruciate Ligament Reconstruction: A Study From the Norwegian Knee Ligament Registry. Am J Sports Med. 2015 Aug;43(8):1902-7. doi: 10.1177/0363546515584041. Epub 2015 May 14. PMID 25977523
- [Background] Jarvinen TL, Sihvonen R, Bhandari M, Sprague S, Malmivaara A, Paavola M, Schunemann HJ, Guyatt GH. Blinded interpretation of study results can feasibly and effectively diminish interpretation bias. J Clin Epidemiol. 2014 Jul;67(7):769-72. doi: 10.1016/j.jclinepi.2013.11.011. Epub 2014 Feb 20. PMID 24560088
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Wideman TH, Finan PH, Edwards RR, Quartana PJ, Buenaver LF, Haythornthwaite JA, Smith MT. Increased sensitivity to physical activity among individuals with knee osteoarthritis: relation to pain outcomes, psychological factors, and responses to quantitative sensory testing. Pain. 2014 Apr;155(4):703-711. doi: 10.1016/j.pain.2013.12.028. Epub 2013 Dec 28. PMID 24378879
- [Background] Ramos-Goni JM, Pinto-Prades JL, Oppe M, Cabases JM, Serrano-Aguilar P, Rivero-Arias O. Valuation and Modeling of EQ-5D-5L Health States Using a Hybrid Approach. Med Care. 2017 Jul;55(7):e51-e58. doi: 10.1097/MLR.0000000000000283. PMID 25521503